CLINICAL TRIAL: NCT05434975
Title: Evaluation of the Effect of Interscalene Block on Intracranial Pressure by Sonographic Measurements of Optic Nerve Sheath Diameter and Internal Jugular Vein Collapsibility Index
Brief Title: The Effect of Interscalene Block on Intracranial Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assistant Professor, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OGundogdu
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Brachial Plexus Block; Intracranial Pressure Increase
Keywords: interscalene brachial plexus block; intracranial pressure; optic nerve sheath diameter; internal jugular vein collapsibility index
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blocked (Experimental): All participants will have single-shot interscalene brachial plexus block with same technique. There is no comparing.
  Interventions: Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — For single shot-ISBP block, 15 ml of 0.5% bupivacaine + 10 ml of 2% prilocaine, a total of 25 ml of local anesthetic, will be administered to all patients.
  For the block procedure, an imaginary horizontal line drawn from the thyroid cartilage to the sternocleidomastoid (SCM) muscle will followed and the lateral of the SCM muscle will be cleaned with povidine iodine. At the C6 level to be blocked, the nerve roots will be detected by ultrasound. 25 ml of local anesthetic will be injected around the plexus roots with a 22 G 80 mm echogenic needle. The distribution of the local anesthetic applied to the area, which expands the tissues and separates the nerve roots from other tissues, will be seen on ultrasound.

SUMMARY:
The study aims to show the effects of interscalene brachial plexus (ISBP) block on intracranial pressure by measuring optic nerve sheath diameter (ONSD) and internal vein collapsibility index (IJV-CI).

DETAILED DESCRIPTION:
40 is the targeted number of patients who are going to have humerus fracture or opened rotator-cuff surgery. Single shot-ISBP block with 25 ml local anesthetic will be performed as anesthetic approach for surgery to all participants. Intraoperative ONSD and IJV-CI measurements will be performed before the ISBP block, 20 minutes and 60 minutes after the block. Hypothesis; external drug-volume effect on internal jugular vein causes decreasing maximum diameter of internal jugular vein (Dmax), venous return from cranium to heart decreases, intracranial pressure can increase.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had elective humeral fracture and open rotator-cuff surgery,
* Patients aged 18-85 years,
* Patients have ASA I-II anesthesia risk according to the American Society of Anesthesiologists (ASA) risk classification,
* Patients that gave consent for participation in the study will be included.

Exclusion Criteria:

* Patients who do not give consent to the study,
* Patients with infection and open wounds in the area of skin puncture and eyelids,
* Patients have any history of intracranial pathology,
* Patients have nerve blockade contraindications such as coagulation disorder and antithrombotic-anticoagulant use,
* Patients have a history of allergy to one of the study drugs,
* Patients have a body mass index over 35 kg/m2,
* Patients with contralateral pneumothorax,
* Patients with severe respiratory distress,
* Patients with uncontrolled hypertension,
* Patients with acute or chronic eye disease,
* Patients with previous eye surgery,
* Patients using a beta-blocker known to increase intraocular pressure,
* Patients using calcium channel blockers, statins and nitrates,
* Patients in need of intraoperative sedation,
* Patients who develope any complications (hoarseness, horner's syndrome, respiratory distress, local anesthetic toxicity) due to ISBP block will be excluded from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter change | Optic nerve sheath diameter will be measured before the block (basal) and it will be measured at 20th and 60th minutes after the block. The change between the measurements of basal and 60th minute and change between basal and 20th minute will be assessed
  Optic nerve sheath diameter will be measured as a unit of millimeter.
Internal jugular vein collapsibility index (IJV-CI) change | IJV-CI will be measured before the block (basal) and it will be measured at 20th and 60th minutes after the block. The change between the measurements of basal and 60th minute, and change between basal and 20th minute will be assessed
  IJV-CI will be measured as a unit of %.
Maximum diameter of internal jugular vein (Dmax) change | Dmax will be measured before the block (basal) and it will be measured at 20th and 60th minutes after the block. The change between the measurements of basal and 60th minute, and change between basal and 20th minute will be assessed
  Dmax will be measured as a unit of millimeter
Minimum diameter of internal jugular vein (Dmin) change | Dmin will be measured before the block (basal) and it will be measured at 20th and 60th minutes after the block. The change between the measurements of basal and 60th minute, and change between basal and 20th minute will be assessed
  Dmin will be measured as a unit of millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Assist. Prof, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No